CLINICAL TRIAL: NCT00076856
Title: A Randomized, Open-Label Phase 2 Study of Temozolomide Added to Whole Brain Radiation Therapy Versus Whole Brain Radiation Therapy Alone for the Treatment of Brain Metastasis From Non-Small Cell Lung Cancer
Brief Title: Temozolomide for Treatment of Brain Metastases From Non-Small Cell Lung Cancer (Study P03247)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03247
Record Dates: First submitted 2004-02-04; First posted 2004-02-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Brain Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: Temozolomide

SUMMARY:
The purpose of this study is to demonstrate improvement in overall survival for the combination of whole brain radiation therapy (WBRT) plus temozolomide (TMZ) versus WBRT alone. Secondary objective is to demonstrate an improvement in the time to radiological CNS progression with the addition of TMZ to WBRT.

ELIGIBILITY:
* Age greater than or equal to 18
* Histologically or cytologically confirmed non-small-cell lung cancer (NSCLC)
* At least one brain metastasis diagnosed within 30 days of randomization
* Brain metastases must not have been previously treated with WBRT or radiosurgery
* No more than 2 sites of extracranial metastases
* May have received prior radiation therapy to the primary tumor and/or systemic metastatic sites
* Meets protocol requirements for specified laboratory values.
* Written informed consent and cooperation of patient
* Appropriate use of effective contraception if of childbearing potential.
* Karnofsky Performance Status KPS greater than 70
* Score less than 2 on all criteria of the Comprehensive Neurological Outcome Scale (CNOS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2004-03-31 (Actual); Primary Completion 2006-03-31 (Actual); Study Completion 2006-03-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival

SECONDARY OUTCOMES:
Time to radiological CNS progression

REFERENCES:
- [Result] Chua D, Krzakowski M, Chouaid C, Pallotta MG, Martinez JI, Gottfried M, Curran W, Throuvalas N. Whole-brain radiation therapy plus concomitant temozolomide for the treatment of brain metastases from non-small-cell lung cancer: a randomized, open-label phase II study. Clin Lung Cancer. 2010 May;11(3):176-81. doi: 10.3816/CLC.2010.n.022. PMID 20439193
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html